CLINICAL TRIAL: NCT03107273
Title: Development of an in Vitro Hematopoietic Culture System and Application to Myelodysplastic Syndromes.
Acronym: HEMASTEM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0035
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hematopoietic Cell Proliferation; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic patient
  Interventions: Other: Dynamic cultures of in vitro hematopoietic stem cells
- Control
  Interventions: Other: Dynamic cultures of in vitro hematopoietic stem cells

INTERVENTIONS:
Other: Dynamic cultures of in vitro hematopoietic stem cells — Improvement of prognostic scores used in myelodysplastic syndromes by identifying by dynamic in vitro culture of hematopoietic stem cells dynamic factors, reflections of ineffective haematopoiesis

SUMMARY:
Myelodysplastic syndromes (MDS) are myeloid hemopathies characterized by ineffective clonal haematopoiesis, peripheral cytopenias and a predisposition to the occurrence of acute myeloid leukemias. Their diagnosis involves a cytological evaluation of the medulla, while their prognosis, in addition to extrinsic factors depending on the patient himself (age, comorbidities), intrinsic factors. The cytological evaluation is subject to a certain subjectivity since qualitative and the diagnosis is sometimes difficult in the absence of marker of clonality. More and more studies emphasize the interest of flow cytometry (CMF) in the diagnosis of SMD: by looking for qualitative and / or quantitative aberrations of the expression of membrane markers, CMF allows to establish scores Diagnosis that we have put in place within the laboratory. However, these studies are based on a static model that studies the phenotypic characteristics of patients at a given time but does not really reflect ineffective hematopoiesis. A dynamic model for in vitro reproduction of hematopoiesis would be an innovative tool for the study of SMD. This project aims to develop and standardize a system of differentiation in liquid medium of hematopoietic stem cells (CSH) in mature cells by studying each stage of the differentiation in terms of proliferation, apoptosis and phenotypic expression. HSCs will be obtained by CD34 + sorting from the medullary sample at diagnosis: the investigator will study cell proliferation, apoptosis and the acquisition of surface markers, in order to identify the quantitative and qualitative abnormalities associated with the differentiation of haematopoietic progenitors Smart. This should make it possible to identify diagnostic and prognostic factors in terms of response to treatment, acutism and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis, major ≥18 years
* Explained in the blood disease department for cytopenia (s)
* For which diagnosis of myelodysplastic syndrome is considered
* Justifying a diagnostic bone marrow (myelogram)
* Having been informed of the progress of this study by the referring physician of the patient during the consultation and having expressed their non-opposition

Exclusion Criteria:

* High-grade myelodysplastic syndromes on IPSS score (intermediate -2 or more) on preliminary cytological analysis
* Acute mesoblastic leukemia from the outset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with anemia and therefore the myelogram finds a low-risk myelodysplastic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Phenotypic aberration detectable in flow cytometry during in vitro erythroid differentiation of hematopoietic stem cells from patients with MDS | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France